CLINICAL TRIAL: NCT05581459
Title: Acute Effects of Muscle Vibration on the Elbow Joint Position Sense in Healthy Young Men
Brief Title: Muscle Vibration and Joint Position Sense
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RRC-2018-007
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Vibration; Exposure
Keywords: Muscle vibration; joint position sense; proprioception; elbow; rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 63 Hz vibration group (Experimental): Vibration of 63 Hz frequency was applied.
  Interventions: Other: 63 Hz Vibration
- 42 Hz vibration group (Active Comparator): Vibration of 42 Hz frequency was applied.
  Interventions: Other: 42 Hz Vibration
- Sham vibration group (Sham Comparator): No actual vibration was applied.
  Interventions: Other: Sham vibration

INTERVENTIONS:
Other: 63 Hz Vibration — Vibrations of 63 Hz were applied with handheld vibration device.
  Arms: 63 Hz vibration group
Other: 42 Hz Vibration — Vibrations of 42 Hz were applied with handheld vibration device.
  Arms: 42 Hz vibration group
Other: Sham vibration — Handheld device was applied to the participants without any vibrations.
  Arms: Sham vibration group

SUMMARY:
The present study aimed to investigate and compare the acute effect of local vibration (63 Hz vs 42 Hz frequencies) on the biceps brachii muscles on the elbow joint position sense (JPS) in healthy young men. Forty-five healthy young men aged 19 to 30 years were enrolled in the study. The participants were randomly assigned to receive either 63 Hz (n=15) or 42 Hz (n=15) or sham vibration (control group) (n=15). Participants in the experimental group received five bouts of 1-minute of each vibration exposure localized to the biceps brachii muscle, with a 1-minute rest between the bouts. Active elbow joint position error (in degrees) was selected as an outcome measure to assess elbow JPS. To measure active elbow joint position error, the subject was made to sit on the chair with eyes closed and shoulders in 0 degree of abduction and elbows fully extended. The examiner passively moved the elbow to 90 degrees of flexion (target position) and maintained it for 10 seconds. The subject was requested to memorize the target position. The subject was asked to actively flex the elbow to the target position from the initial starting position (elbow fully extended) and hold it for 5 seconds. Three trials were conducted, with a 30-second rest given between each trial. The target and reproduced angles in each trial were measured using a standard plastic goniometer. The difference between the target and reproduced angles in each trial was calculated to determine active elbow joint position error. Measurements were taken at baseline and immediately after the vibration protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young men

Exclusion Criteria:

* history of recent upper extremity surgery
* history of sensory deficits in the upper extremity
* recent upper extremity injury
* undergoing any resistance training

Ages: 19 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Active elbow joint position error | 1 day
  Participants were asked to actively reproduce a target position of the elbow joint.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No